CLINICAL TRIAL: NCT02257749
Title: Comparing Active Rehabilitation to a Comprehensive Education Intervention for Youth With Persistent Post-concussion Symptoms Following Concussion.
Brief Title: Trial Study of an Exercise Program for Youth With Persistent Symptoms After Concussion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility; challenges with recruitment
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-459
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Concussion; Sport-Related Concussion; Mild Traumatic Brain Injury
Keywords: Concussion; Persistent Symptoms; Children; Exercise; Adolescents; Active Rehabilitation; Education
MeSH Terms: conditions — Brain Concussion; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Rehabilitation (Experimental): Active Rehabilitation Intervention and Comprehensive Education Intervention (Standard Care)
  Interventions: Other: Active Rehabilitation; Other: Comprehensive Education Intervention (Standard Care)
- Comprehensive Education Intervention (Active Comparator): Comprehensive Education Intervention (Standard Care) only
  Interventions: Other: Comprehensive Education Intervention (Standard Care)

INTERVENTIONS:
Other: Active Rehabilitation — The active rehabilitation intervention is a 6-week graded rehabilitation program, consisting of four components that are anchored in neuroscience evidence.The four components include: 1) aerobic exercise 2) coordination exercise 3) visualization 4) home program.
  Arms: Active Rehabilitation
Other: Comprehensive Education Intervention (Standard Care) — An initial education session will be provided by an occupational therapist related to general concussion information and outcomes, as well as strategies for symptom management following concussion.

SUMMARY:
The purpose of this randomized control trial study is to determine if an active rehabilitation (low intensity exercise program) in combination with a comprehensive education intervention (standard care) is more effective than the comprehensive education intervention alone in reducing post-concussion symptoms and improving participation in daily activities in youth who have persistent post-concussion symptoms.

DETAILED DESCRIPTION:
There is a portion of youth who continue to experience persistent post-concussion symptoms beyond the first few weeks of injury. There is limited evidence with respect to the best ways to treat persistent post-concussion symptoms in youth following concussion. There is a small amount of literature that suggests active rehabilitation as a positive intervention for promotion of recovery of persistent post-concussion symptoms. However, this approach to rehabilitation has yet to be explored using a randomized control trial protocol.

Therefore, this study aims to answer the following question: Is a 6 week active rehabilitation program in combination with a comprehensive education intervention (standard care) effective in reducing post-concussive symptoms and improving functional recovery compared to receiving comprehensive education intervention alone among youth experiencing persistent post-concussion symptoms?

We hypothesize:

1. youth ages 10 to 18 years who present with persistent self-reported post-concussion symptoms 4 weeks after the initial injury and receive the active rehabilitation intervention, will present with decreased post-concussion symptoms at the completion of the intervention.
2. youth ages 10 to 18 years who receive the active rehabilitation intervention, will present with more complete functional recovery and increased participation in unrestricted physical activity at the completion of the active rehabilitation intervention compared to children receiving the comprehensive education intervention only

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of concussion
* have at least one post-concussion symptom (as measured by the Post Concussion Symptom Inventory)
* are at least 4 weeks post injury
* between the ages of 10 and 18 years
* ability to speak English
* ability to demonstrate capacity to consent to study

Exclusion Criteria:

* prior moderate or severe brain injury
* neck pain/dysfunction or oculormotor/vestibular dysfunction, developmental delays, mental health disorders or chronic pain conditions that prevent participation in active rehabilitation, assessment of gait and balance, or participation in cognitive testing
* participating in any other physical rehabilitation interventions for post-concussion symptoms (e.g., physiotherapy, massage therapy, chiropractic) at time of enrollment and throughout the duration of the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Post-Concussion Symptoms | Week 0 (Baseline)
  The Post-Concussion Symptom Inventory will be used. This is a self report questionnaire that asks about subjectively experienced symptoms (presence and severity) such as headache, dizziness, memory troubles, after concussion.
Post Concussion Symptoms | Week 2
  The Post-Concussion Symptom Inventory will be used. This is a self report questionnaire that asks about subjectively experienced symptoms (presence and severity) such as headache, dizziness, memory troubles, after concussion.
Post Concussion Symptoms | Week 6 (upon completion of intervention)
  The Post-Concussion Symptom Inventory will be used. This is a self report questionnaire that asks about subjectively experienced symptoms (presence and severity) such as headache, dizziness, memory troubles, after concussion.

SECONDARY OUTCOMES:
Mood | Week 0 (Baseline)
  The Beck Depression Inventory for Youth- Second Edition will be used. This is a screen that was designed for youth and provides insight into negative thoughts and feelings towards self, life and future.
Mood | Week 6 (upon completion of the intervention)
  The Beck Depression Inventory for Youth- Second Edition will be used. This is a screen that was designed for youth and provides insight into negative thoughts and feelings towards self, life and future.
Behavior | Week 0 (Baseline)
  The Child Behavior Checklist will be used. It is designed to identify emotional and behavioral concerns in youth.
Behavior | Week 6 (upon completion of the intervention)
  The Child Behavior Checklist will be used. It is designed to identify emotional and behavioral concerns in youth.
Energy Level | Week 0 (Baseline)
  Pediatric Quality of Life Multidimensional Fatigue Scale will be used to examine fatigue
Energy Level | Week 6 (upon completion of the intervention)
  Pediatric Quality of Life Multidimensional Fatigue Scale will be used to examine fatigue
Quality of Life Level | Week 0 (Baseline)
  Pediatric Quality of Life Generic Module will be used to look at quality of life
Quality of Life Level | Week 6 (upon completion of the intervention)
  Pediatric Quality of Life Generic Module will be used to look at quality of life
SCAT Balance | Week 0 (Baseline)
  Sport Concussion Assessment Tool- 3rd Edition Balance Subtest will be used. This measure looks at static balance and postural stability. Youth are asked to perform three different stances on a firm surface for 20 seconds each.
Balance | Week 0 (Baseline)
  Bruininks-Oseretsky Test of Motor Proficiency, Second Edition Balance Subtest will be used. This is used to assess static and dynamic balance with focus on the youth's anticipatory postural control.
Balance | Week 6 (upon completion of the intervention)
  Bruininks-Oseretsky Test of Motor Proficiency, Second Edition Balance Subtest will be used. This is used to assess static and dynamic balance with focus on the youth's anticipatory postural control.
Neurocognitive | Week 0 (Baseline)
  ImPACT testing will be done. This is a computer based program designed to assess multiple aspects of cognitive functioning following a concussion.
Neurocognitive | Week 6 (upon completion of the intervention)
  ImPACT testing will be done. This is a computer based program designed to assess multiple aspects of cognitive functioning following a concussion.
Anxiety | Week 0 (Baseline)
  State Trait Anxiety Scale will be used to look at parental anxiety
Anxiety | Week 6 (upon completion of the intervention)
  State Trait Anxiety Scale will be used to look at parental anxiety
Activity Participation | Week 0 (Baseline)
  Physical Activity Questionnaire for Children and Adolescents will be used to look at the physical activities performed in the 7 days prior to evaluation.
Satisfaction Level | Week 0 (Baseline)
  Pediatric Quality of Life Health Care Satisfaction Generic Module will be used to gain an understanding of the participants' perceptions of the quality and effectiveness of the intervention.
Acute Concussion Evaluation | Week 0 (Baseline)
  Acute Concussion Evaluation will be used to collect demographic information such as characteristics of the injury, signs and symptoms of the injury, and risk factors that may predict prolonged recovery.
Occupational Performance | Week 0 (Baseline)
  The Canadian Occupational Performance Measure will be used to identify occupational performance issues as a platform for goal setting. Participants' rate their satisfaction and performance in self-identified activities that they would like to improve their satisfaction and performance in.
Occupational Performance | Week 6 (upon completion of the intervention)
  Participants re-rate their satisfaction and performance in the three areas they self-identified as occupational concerns at week 0 (baseline)
Balance | Week 6 (upon completion of intervention)
  Sport Concussion Assessment Tool- 3rd Edition Balance Subtest will be used. This measure looks at static balance and postural stability. Youth are asked to perform three different stances on a firm surface for 20 seconds each.
Activity Participation | Week 6 (upon completion of the intervention)
  Physical Activity Questionnaire for Children and Adolescents will be used to look at the physical activities performed in the 7 days prior to evaluation.
Activity Participation | Week 2
  Physical Activity Questionnaire for Children and Adolescents will be used to look at the physical activities performed in the 7 days prior to evaluation.
Satisfaction Level | Week 6 (upon completion of the intervention)
  Pediatric Quality of Life Health Care Satisfaction Generic Module will be used to gain an understanding of the participants' perceptions of the quality and effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Reed, PhD, MSc(OT), Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital/ Bloorview Research Institute
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Reed N, Greenspoon D, Iverson GL, DeMatteo C, Fait P, Gauvin-Lepage J, Hunt A, Gagnon IJ. Management of persistent postconcussion symptoms in youth: a randomised control trial protocol. BMJ Open. 2015 Jul 31;5(7):e008468. doi: 10.1136/bmjopen-2015-008468. PMID 26231756